CLINICAL TRIAL: NCT03549897
Title: A Randomized, Single-Dose, Double-Blind, Double-Dummy, Four-Period, Four-Sequence, Four-Treatment, Placebo and Active Controlled, Comparative, Multiple-Center, Crossover-Design, Bronchoprovocation Study to Evaluate the Pharmacodynamic Equivalence of Albuterol Sulfate Inhalation Aerosol, eq 90 mcg Base (Amneal Ireland Limited) to PROAIR® HFA (Albuterol Sulfate) Inhalation Aerosol, eq 90 mcg Base (Teva Respiratory, LLC) in Patients With Stable, Mild Asthma
Brief Title: Bronchoprovocation Study to Evaluate the Pharmacodynamics of Albuterol Sulfate Inhalation Aerosol, eq 90 mcg Base
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amneal Ireland Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AI-ABL-001
Record Dates: First submitted 2018-04-06; First posted 2018-06-08 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo Product (Placebo Comparator): One actuation each from two different placebo Reference inhalation aerosols and one actuation each from two different placebo Test inhalation aerosols
  Interventions: Drug: Placebo
- 90 mcg Reference Product (Active Comparator): One actuation each from the Reference inhalation aerosol and the placebo Reference inhalation aerosol and one actuation each from two different placebo Test inhalation aerosols
  Interventions: Drug: 90 mcg Reference Product
- 180 mcg Reference Product (Active Comparator): One actuation each from two different Reference inhalation aerosol and one actuation each from two different placebo Test inhalation aerosols
  Interventions: Drug: 180 mcg Reference Product
- 90 mcg Test Product (Experimental): One actuation each from the Test inhalation aerosol and the placebo Test inhalation aerosol and one actuation each from two different placebo Reference inhalation aerosols
  Interventions: Drug: 90 mcg Test Product

INTERVENTIONS:
Drug: Placebo — Placebo Product
  Arms: Placebo Product
Drug: 90 mcg Reference Product — 90 mcg Reference Product - PROAIR HFA ALBUTEROL SULFATE [TEVA RESPIRATORY, LLC]
  Other Names: Albuterol
  Arms: 90 mcg Reference Product
Drug: 180 mcg Reference Product — 180 mcg Reference Product- PROAIR HFA ALBUTEROL SULFATE [TEVA RESPIRATORY, LLC]
  Other Names: Albuterol
  Arms: 180 mcg Reference Product
Drug: 90 mcg Test Product — 90 mcg Test Product - ALBUTEROL SULFATE HFA [AMNEAL IRELAND LIMITED]
  Other Names: Albuterol
  Arms: 90 mcg Test Product

SUMMARY:
This randomized, single-dose, double-blind, double-dummy, four-period, four-sequence, four-treatment, placebo and active controlled, comparative, multiple-center, crossover-design bronchoprovocation study has been designed to evaluate the pharmacodynamic equivalence of albuterol sulfate HFA inhalation aerosol, eq 90 mcg base (Amneal Ireland Limited) to PROAIR® HFA (albuterol sulfate) Inhalation Aerosol, eq 90 mcg base (Teva Respiratory, LLC) in patients with stable mild asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female subjects (18-65 years of age).
* Stable mild asthmatics based on National Asthma Education and Prevention Program (NAEPP) guidelines.
* FEV1 ≥ 80% of predicted.
* Airway responsiveness to methacholine demonstrated by a pre-albuterol-dose (baseline) PC20 ≤ 8 mg/mL.
* Nonsmokers for at least six months prior to the study and a maximum smoking history of five pack-years (the equivalent of one pack per day for five years).
* Written informed consent

Exclusion Criteria:

* Evidence of upper or lower respiratory tract infection (e.g., pneumonia, bronchitis, sinusitis) within six weeks prior to the study.
* History of seasonal asthma exacerbations, in which case the subject should be studied outside of the relevant allergen season.
* History of cystic fibrosis, bronchiectasis or other respiratory diseases.
* History of cardiovascular, renal, neurologic, liver or endocrine dysfunction, including ECG with evidence of ischemic heart disease.
* Treatment in an emergency room or hospitalization for acute asthmatic symptoms or need for daily oral corticosteroids within past three months.
* Known intolerance or hypersensitivity to any component of the albuterol MDI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Primary Pharmacodynamic Endpoint Post-dose PC20 | 6 weeks
  Provocative concentration of the methacholine challenge agent required to reduce the FEV1 by 20% following administration of differing doses of albuterol or placebo by inhalation. The 20% reduction in FEV1 will be determined relative to the post-saline FEV1 measure before the placebo or albuterol administration.

CONTACTS AND LOCATIONS:
Overall Officials: Irshad Haque, Study Director — Amneal Pharmaceuticals, LLC
Locations (1):
- Amneal Pharmaceuticals LLC, Brookhaven, New York, United States

IPD SHARING:
Plan to Share IPD: No